CLINICAL TRIAL: NCT01256866
Title: Sedation of Mechanically Ventilated Critically Ill Patients: Midazolam Versus Dexmedetomidine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Ethics Committee, Hospital Sao Domingos
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: hsd130947
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-11

CONDITIONS: Mechanically Ventilated Patients; Sedation; Dexmedetomidine; Midazolam
Keywords: Dexmedetomidine; Midazolam; Sedation; Mechanical ventilation; Critically ill patients
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DEXMEDETOMIDINE, SEDATION (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- Midazolam, sedation, (Active Comparator)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: DEXMEDETOMIDINE, SEDATION
Drug: Midazolam
  Arms: Midazolam, sedation,

SUMMARY:
The aim of this prospective randomized study is to compare the safety and efficacy of two strategies for sedation of critically ill patients submitted to mechanical ventilation: continuous intravenous infusion of dexmedetomidine versus intravenous bolus of midazolam. The two groups will be compared as to the incidence of of delirium, evaluated with the Confusion Assessment Method for ICU (CAM-ICU) and the percentage of time within the target sedation using the Richmond Agitation-Sedation Scale (RAAS).Eligible patients will be 18 years or older intubated and mechanically ventilated for less than 48 hours prior to start of study drug and anticipated ventilation duration of at least 48 hours. Calculated sample size is 146 patients (73 patients in each group)

ELIGIBILITY:
Inclusion Criteria:

* Adult mechanically ventilated, critically ill patients

Exclusion Criteria:

* pregnancy or lactation, severe liver disease, hearth rate less than 50, hypotension despite volemic repletion and vasoactive drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-10 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium

SECONDARY OUTCOMES:
PERCENTAGE OF TIME WITHIN THE TARGET SEDATION

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sao Domingos, São Luís, Maranhão, Brazil